CLINICAL TRIAL: NCT06358638
Title: Sickle Cell Disease Transplant Using a Nonmyeloablative Approach: Adding Daratumumab for Patients With Anti-donor Red Cell AntibodY
Brief Title: Sickle Cell Disease Transplant Using a Nonmyeloablative Approach for Patients With Anti-donor Red Cell Antibody
Acronym: SUN-RAY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: Alberta Children's Hospital (Other); The Hospital for Sick Children (Other); Levine Children's Hospital (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Nationwide Children's Hospital (Other); Children's Hospital at Montefiore (Other); Doris Duke Charitable Foundation (Other); Janssen Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Robert Nickel, MD, Children's National Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000859
Record Dates: First submitted 2024-04-02; First posted 2024-04-10 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; ABO Mismatch; SUN-RAY; Matched Sibling Donor (MSD)
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — daratumumab; Alemtuzumab; Sirolimus; Whole-Body Irradiation

STUDY DESIGN:
Intervention Model Description: Sickle cell patients, who have matched sibling donors with anti-donor RBC antibodies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Recipients with a major ABO incompatible donor (Experimental): Patients in this cohort are treated pre-HCT with Daratumumab, intravenously, on days -49, -42, -35 and -28. The conditioning regimen will consist of alemtuzumab, given subcutaneously, daily for 5 days (days -7 to -3) and low dose total body irradiation (TBI) 300 cGY on day -2 with gonadal shielding. Sirolimus will be given as GVHD prophylaxis for the first year with weaning thereafter based on donor T-cell chimerism. G-CSF, at 5 mcg/kg/day, will be given post stem cell infusion until neutrophil engraftment is achieved.
  Interventions: Drug: Daratumumab; Drug: Alemtuzumab; Drug: Sirolimus; Radiation: Total Body Irradiation
- Recipients with red cell alloantibodies (non-ABO) against donor antigens (Experimental): Patients in this cohort are treated pre-HCT with Daratumumab, intravenously, on days -49, -42, -35 and -28. The conditioning regimen will consist of alemtuzumab, given subcutaneously, daily for 5 days (days -7 to -3) and low dose total body irradiation (TBI) 300 cGY on day -2 with gonadal shielding. Sirolimus will be given as GVHD prophylaxis for the first year with weaning thereafter based on donor T-cell chimerism. G-CSF, at 5 mcg/kg/day, will be given post stem cell infusion until neutrophil engraftment is achieved.
  Interventions: Drug: Daratumumab; Drug: Alemtuzumab; Drug: Sirolimus; Radiation: Total Body Irradiation

INTERVENTIONS:
Drug: Daratumumab — Daratumumab is a cytotoxic monoclonal antibody (IgG1k) to CD38 and is commercially approved to treat multiple myeloma. CD38 is expressed on several types of blood cells including B-cells, antibody-secreting plasma blasts and plasma cells. As a result, it has been used to treat antibody-mediated diseases, including children with antibody-mediated cytopenias post-HCT.
  Other Names: Darzalex
Drug: Alemtuzumab — Alemtuzumab is a humanized monoclonal antibody specific to lymphocyte antigens. It is a recombinant DNA-derived humanized monoclonal antibody (Campath-1H) that is directed against the 21-28 kD cell surface glycoprotein, CD52.
  Other Names: Campath-1H
Drug: Sirolimus — Sirolimus is an mTOR inhibitor immunosuppressant used to prevent organ transplant rejections as well as treat lymphangioleiomyomatosis and adults with perivascular epithelioid cell tumors.
  Other Names: Rapamune
Radiation: Total Body Irradiation — Total body irradiation is a form of radiotherapy used primarily as part of the preparative regimen for haematopoietic stem cell transplantation. The radiation is given in a low dose so that normal tissues can repair themselves.
  Other Names: TBI

SUMMARY:
This multicenter prospective study seeks to determine if daratumumab given, prior to HLA-identical sibling donor transplantation using alemtuzumab, low dose total-body irradiation, and sirolimus, can prevent pure red blood cell aplasia with an acceptable safety profile in patients with anti-donor red blood cell antibodies, achieving an event-free survival similar to transplanted patients without such antibodies.

DETAILED DESCRIPTION:
This study addresses an important question: Can daratumumab safely be administered prior to matched sibling donor (MSD) nonmyeloablative hematopoietic cell transplant (HCT) for SCD to avoid pure red blood cell aplasia in patients at risk of this complication? and thus achieve an event-free survival similar to patients without anti-donor red blood cell (RBC) antibodies?

Patients with anti-donor RBC antibodies, which includes patients with major ABO mismatch and other RBC alloantibodies against donor, have largely been excluded from the nonmyeloablative HCT approach given their risk of delayed donor RBC engraftment and/or hemolysis post-HCT. Exclusion of these patients limits access to less toxic curative therapies for this population at risk for toxicity due to their underlying multisystem disease. To address this need, we propose a multicenter clinical trial of Sickle cell disease Using a Nonmyeloablative approach: adding daratumumab for patients with anti-donor Red cell AntibodY (SUN-RAY). If successful, this trial will increase access to MSD nonmyeloablative HCT in SCD and will provide important safety and efficacy data for the use of daratumumab in the pre-HCT setting as well as in patients with SCD who have limited RBC donor options due to alloimmunization.

This is a phase 2 study given that the studied nonmyeloablative conditioning backbone (alemtuzumab, 300 cGY TBI, sirolimus) has been previously used effectively in both adults and children with SCD. Daratumumab will be added to this backbone with a washout period of 4 weeks prior to HCT infusion. Small case series have demonstrated that daratumumab is well tolerated either pre-HCT to treat patients with antibodies against mismatched donor HLA antigens, or post-HCT in patients with autoimmune cytopenias. The experience of the phase 2 clinical trial NCT03384654 studying daratumumab in pediatric acute lymphoblastic leukemia provides additional support for the safety and dosing of daratumumab for this study.

ELIGIBILITY:
Inclusion Criteria:

General:

* Patients with SCD age 2-24.99 years who have a healthy HLA-identical sibling donor with major ABO incompatibility OR patients with RBC alloantibodies against other donor RBC antigens.
* Patients must have an absolute neutrophil count of 1 x 109/L and a platelet count of 100 x 109/L.
* Lansky/Karnofsky score of, at least, 70.

Patients with genotypes hemoglobin SS and Sβ0 thalassemia must have at least one of the following:

* History of an abnormal transcranial Doppler measurement defined as TCD velocity ≥200 cm/sec by the non-imaging technique measured at a minimum of two separate occasions.
* Progression of CNS vasculopathy on MRA determined to be secondary to SCD.
* History of cerebral infarction on brain MRI (overt stroke, or silent stroke if ≥3 mm in one dimension, visible in two planes on fluid-attenuated inversion recovery T2-weighted images).
* History of two or more episodes of Acute Chest Syndrome (ACS) in lifetime.
* History of three or more SCD pain events requiring treatment with an opiate or IV pain medication in lifetime.
* History of any hospitalization for a complication secondary to SCD (does NOT include empiric hospitalizations for fever only).
* History of two or more episodes of priapism.
* Administration of regular RBC transfusions (≥8 transfusions episodes in the previous 12 months).
* At least two episodes of splenic sequestration requiring red blood cell transfusion or splenectomy after at least one episode of splenic sequestration.

Patients with all other sickle genotypes (e.g. hemoglobin SC, Sβ+ thalassemia, etc.) must have at least one of the following:

* Clinically significant neurologic event (overt stroke).
* History of two or more episodes of ACS in the 2-year period preceding enrollment.
* History of three or more SCD pain events requiring treatment with an opiate or IV pain medication (inpatient or outpatient) in the 1-year period preceding enrollment.
* History of any hospitalization for SCD pain or ACS while receiving hydroxyurea treatment.
* History of two or more episodes of priapism (erection lasting ≥4 hours or requiring emergent medical care).
* Administration of regular RBC transfusions (≥8 transfusions in the previous 12 months)
* At least two episodes of splenic sequestration requiring red blood cell transfusion or splenectomy after at least one episode of splenic sequestration.

Exclusion Criteria:

* Life expectancy less than 6 month
* Pregnant or breastfeeding patients.
* Infectious Disease: Uncontrolled bacterial, viral or fungal infections (undergoing appropriate treatment and with progression of clinical symptoms) within 1 month prior to conditioning. Patients with febrile illness or suspected minor infection should await clinical resolution prior to starting conditioning. Patients with confirmed seropositivity for HIV and patients with active or resolved Hepatitis B or C determined by serology and/or NAAT are excluded.
* Liver: Direct (conjugated) bilirubin > 1.5 mg/dL. Transaminases >5x upper limit of normal for age.
* Cardiac: Left ventricular shortening fraction <25% or ejection fraction <50% by ECHO. Uncontrolled cardiac arrhythmia.
* Kidney: Estimated creatinine clearance less than 60 mL/min/1.73m2.
* Pulmonary function: Diffusion capacity of carbon monoxide (DLCO) <35% (adjusted for hemoglobin). Baseline oxygen saturation <94% at rest or PaO2 <70. Known moderate or severe persistent asthma within the past 2 years, or uncontrolled asthma of any classification.
* Heme: Available, medically suitable, and equivalent HLA-matched sibling donor, who does not have major ABO incompatibility or express RBC antigens against which the patient is alloimmunized.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2044-09 (Estimated); Study Completion 2054-09 (Estimated)

PRIMARY OUTCOMES:
To determine the event-free survival of children and adolescents with SCD undergoing nonmyeloablative HCT who received 4 doses of pre-HCT daratumumab for donor-directed red blood cell antibodies. | 1-year post-transplant
  Event-free survival rate at 1 year with events including death, graft failure (donor myeloid chimerism <10% or second HCT), grade II-IV GVHD, and serious pure red blood cell aplasia (persistent reticulocytopenia and need for red blood cell transfusion support after day +100).

SECONDARY OUTCOMES:
To evaluate changes in antibodies to red blood cell antigens pre and post exposure to daratumumab and HCT. | 100 days post-transplant
  Antibodies titers against donor red blood cell antigens pre and post exposure to daratumumab. Anti-A and Anti-B titers, RBC alloantibody testing at baseline, day -7, day 0, day +30, and day +100.
To characterize the safety of adding pre-HCT daratumumab to the conditioning regimen, as defined by adverse events grade 3 or greater. | 1-year post-transplant
  Proportion of patients with infusion reactions and grade 3 adverse events related to daratumumab, and infections requiring treatment in the first year post-HCT, with comparison to historical controls on the SUN study.

OTHER OUTCOMES:
To compare alemtuzumab levels, in mcg/mL, post-HCT among patients treated with daratumumab, with patients not treated with daratumumab on the SUN study. | Through end of study
  Testing alemtuzumab levels on day 0, +7, +14 and +30.
To compare immune reconstitution among patients treated with daratumumab, with patients not treated with daratumumab on the SUN study. | Through end of study
  Testing immune cell subsets at day +180 and +365.
To compare donor chimerism (lymphoid vs myeloid) post-HCT among patients treated with daratumumab, with patients not treated with daratumumab on the SUN study. | Through end of study
  Testing donor chimerism at day +30, +60, +100, +150, +180, +270 and +365.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Nickel, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No